## Clinical Study of Intradialytic Combined Exercise Program Constructed by Systematic Review in Maintenance Hemodialysis Patients

Ethics Committee Approval (No 2018538)

Investgator Mei Huang

Edited on November 10, 2018

## Informed consent forms

Dear participant:

Hello!

The study would conduct by Mei Huang, a graduate student of the Department of Nursing, Xi'an Jiaotong University, and under the supervision and guidance of the tutor Aili Lv. The aim of this study is to understand the effects of exercise programs which was conducted by investigators' former systematic review on dialysis efficacy, physical function, physiological indicators and quality of life in maintenance hemodialysis patients, and provide scientific and feasible exercise program for maintenance hemodialysis patients and clinical staff.

We will provide you with relevant knowledge of sports during the hemodialysis, and give you professional guidance and supervision. We will provide you with the appropriate exercise intensity and exercise volume according to your own physical condition. If you feel any discomfort during exercise, you can stop exercise immediately and communicate with the investigator, doctors or nurses of the blood purification center.

We will also need you to fill out a questionnaire about health-related quality of life before exercise intervention, at the end of 12 weeks and 24 weeks of exercise. And we will test your physical function to evaluate the effects of exercise.

This research needs your support and cooperation, please rest assured:

- 1. This study won't cause any physical or mental harm to you and your family.
  - 2. You will not be charged any fees throughout the study.
- 3. This study requires patients to participate fully in the process. You can choose whether or not to participate in the study based on your specific circumstances and family opinions. Even if you have signed an informed consent form, you still have the right to withdraw from the study without any impact on you.
  - 4. We will keep the information you provide confidential.

## Consent Form

I agree to participate in the above study, and the investigator explained to me that the purpose of the study has been understood, and even if I have signed this consent, I still have the right to withdraw from the study without any impact on my medical services and treatment. The information obtained is for research use only and will be kept strictly confidential.

Thank you very much for your understanding, support and help!

| J | 3 | υ, | 11 | 1 |
|---|---|---|---|---|
| Researcher's signature: Patient signature: | | | | |
| | Date: | year | month _ | day |